CLINICAL TRIAL: NCT01364805
Title: Translation of in Vitro and in Vivo Ascorbate Research Into a New Treatment Option for Pancreatic Cancer: Phase I/IIa Clinical Trial
Brief Title: New Treatment Option for Pancreatic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Jeanne Drisko, MD, CNS, FACN (Other)
Collaborators: Lotte & John Hecht Memorial Foundation (Other); University of Kansas Medical Center (Other)
Responsible Party: Sponsor-Investigator, Jeanne Drisko, MD, CNS, FACN, Director Integrative Medicine, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12505
Record Dates: First submitted 2011-05-24; First posted 2011-06-02 (Estimated); Last update posted 2018-06-19 (Actual); Status verified 2018-06

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Ascorbic Acid; Gemcitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- PK Intravenous Vitamin C and Gemcitabine (Experimental): Week 1: 2 visits for escalating doses of intravenous ascorbic acid (IV C). First dose 25 gm followed by 50 gm 2nd visit. Week 2: 3 visits escalating doses of IV C, 75 grams, 100 grams, and 125 grams. Week 3: 2 visits pharmacokinetic evaluation of intravenous ascorbic acid alone at 125 grams; return to the infusion clinic the following morning for a 24 hour blood draw; 2nd visit receive the first infusion of gemcitabine chemotherapy for PK evaluation of gemcitabine alone. Week-4: gemcitabine and IV C co-administered for pharmacokinetics of both drugs to assess for PK variability related to drug-drug interactions. Subjects will return to the infusion clinic the following morning for 24 hour blood draw.
  Interventions: Drug: Intravenous Vitamin C; Drug: Gemcitabine

INTERVENTIONS:
Drug: Intravenous Vitamin C — The first 5 study visits will all take place in the General Clinical Research Center (GCRC). During these visits you will receive IV doses of Vitamin C. The dose of Vitamin C will be started at 25 grams and may be increased up to 125 grams over a two week period. There may be changes in the amount of Vitamin C that you receive based on your blood test levels. The study staff will go over this in more detail with you. The amount of fluid you receive depends on the dose and can be from 2 1/3 cups to 5 cups.
  Other Names: IV ascorbic acid
Drug: Gemcitabine — Participants receive dexamethasone 10 mg as pretreatment antiemetic; may be given ondansetron, granisetron, or dolasetron, per oncologist. Gemcitibane 1,000mg/m2 IV over 30 minutes Q 21 days. Cycle of treatment: infusions once weekly for 2 consecutive weeks followed by 1 week of rest to continue treatment schedule until they experience disease progression or unacceptable toxicity. CR, PR or SD: treatment will be continued for at least 6 cycles. Discontinuation of therapy may be considered if agreed upon by the participant and oncologist. Dose Modifications: If the patient experiences more than one toxicity, each requiring a dose reduction, follow the guidelines that give the largest dose reduction for the drug. Subsequent doses can be adjusted to as low as 500 mg/m2 for gemcitabine.
  Other Names: Gemsar

SUMMARY:
In the United States, approximately 30,000 new cases of pancreatic cancer are diagnosed each year and an almost equal number of deaths are related to this cancer. Different types of chemotherapeutic treatments are used that target different parts of the cancer cell with some success, but there is room for other treatment options.

It is known that people with cancer are using high doses of intravenous vitamin C also known as ascorbate, as a cancer treatment and this is occurring frequently. When Vitamin C is given in this manner, it is not taken by mouth; instead, it enters your body through an IV (intravenous) site, or tube that is inserted through a needle into your vein. If you have a port-a-cath in place, the IV will be given using your port. When Vitamin C enters your body through an IV site, it is known that it acts like a drug and not a vitamin. It produces a substance around the cancer cells called hydrogen peroxide. It has been seen in animal research studies that hydrogen peroxide kills the cancer cells while leaving the normal cells unharmed.

Currently the FDA does not approve the use of high-dose intravenous Vitamin C as a cancer treatment. The use of intravenous Vitamin C in this study is experimental. Furthermore, it is important to know that we do not expect the intravenous Vitamin C given in this study to be healing for the treatment of your cancer.

DETAILED DESCRIPTION:
The purpose of this study is to determine if it is safe to give Vitamin C by the vein at high doses to people with pancreatic cancer and if Vitamin C interferes with how well the chemotherapy works on cancer cells. This study will also look at how the body processes of Vitamin C. This study will also help researchers to learn more about long Vitamin C stays in the blood stream, and how rapidly it is used by the body.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be 21 years of age or older and have histologically or cytologically diagnosed carcinoma of the pancreas defined as locally advanced or metastatic and if locally advanced, not eligible for surgical resection
* The patient must screened for eligibility and have care approved by treating oncologist; the oncology care is to be dictated by the oncology team and patient and will include gemcitabine chemotherapy.
* ECOG Performance Status 0-2 Eastern Cooperative Oncology Group Performance Status Grade 0 = Fully active, able to carry on all pre-disease activities without restriction Grade 1= Restricted in physical strenuous activity but ambulatory and able to carry out work of a light or sedentary nature e.g. light housework, office work Grade 2 = Ambulatory and capable of all self care but unable to carry out any work activities, up and about more than 50% of waking hours
* Laboratory: ANC ≥1,500/mm3, Hemoglobin > 8g/dL, platelet ≥ 1000,000/mm3, total bilirubin ≤ 1.5 mg/dL (in the absence of neoplastic involvement), creatinine ≤2.0 mg/dL, transaminase (AST/ALT) ≤2.5X upper limit, urine uric acid < 1,000mg/d, urine pH <6, urine oxalate <60 mg/d.
* Patients who have no language barrier, are cooperative, and can give informed consent before entering the study after being informed of the medications and procedures to be used in this study may participate.

Exclusion Criteria:

* Glucose-6-phosphate-dehydrogenase (G6PD) deficiency
* History of oxalate renal calculi; urine oxalate level > 60 mg/d at baseline
* History of bleeding disorder, iron overload or hemochromatosis
* Prior chemotherapy or currently receiving chemotherapy or radiation therapy or enrolled in other trials currently or in the preceding 1 month.
* Patients with evidence of a significant psychiatric disorder by history/examination that would prevent completion of the study will not be allowed to participate.
* ECOG Performance Status of 3-4. Grade 3 = capable of only limited self care, confined to bed or chair more than 50% of waking hours. Grade 4 = completely disabled. Cannot carry on any self care. Totally confined to bed or chair.)
* Co-morbid condition that would affect survival: end stage congestive heart failure, unstable angina, myocardial infarction within 6 weeks of study, uncontrolled blood sugars ≥ 300 mg/dL, patients with known chronic active hepatitis or cirrhosis.
* Patients who consume an excess of alcohol or abuse drugs (an excess of alcohol is defined as more than four of any one of the following per day: 30mL distilled spirits, 340mL beer, or 120mL wine) will not be allowed.
* Patients who smoke tobacco products will not be allowed to participate.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2011-04; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Determine safety of combined gemcitabine chemotherapy with IV ascorbate. | 12 months
  This will be accomplished by enrolling up to 14 participants fitting inclusion criteria into the Phase I portion of the trial: 7 participants will be enrolled at the determined dose levels and if no significant adverse event is identified, then 7 additional participants will be enrolled. Safety will be assessed by obtaining the following evaluations: toxicity graded by the NCI CTCAE v 4.0, urinalysis pre- and post-infusion, ECG, basic metabolic panel, bicarbonate (pH surrogate marker), CBC, and osmolality.

SECONDARY OUTCOMES:
Assess pharmacokinetic and pharmacodynamic interactions when adding IV AA to front-line gemcitabine chemotherapy in the treatment of locally advanced or metastatic pancreatic cancer not eligible for surgical resection. | 12 months
  By measuring PK data when combining gemcitabine chemotherapy along with IV ascorbate on the same day, it will be determined if there are reduced gemcitabine levels in the presence of ascorbate. Initially 7 participants will be enrolled and if no significant interaction defined, an additional 7 will be enrolled.

CONTACTS AND LOCATIONS:
Overall Officials: Jeanne Drisko, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Kansas, United States

REFERENCES:
- [Result] Polireddy K, Dong R, Reed G, Yu J, Chen P, Williamson S, Violet PC, Pessetto Z, Godwin AK, Fan F, Levine M, Drisko JA, Chen Q. High Dose Parenteral Ascorbate Inhibited Pancreatic Cancer Growth and Metastasis: Mechanisms and a Phase I/IIa study. Sci Rep. 2017 Dec 7;7(1):17188. doi: 10.1038/s41598-017-17568-8. PMID 29215048